CLINICAL TRIAL: NCT00413062
Title: A Randomized, Open-Label, Comparative, Multi -Center Trial to Evaluate Contraceptive Efficacy, Cycle Control, Safety and Acceptability of a Monophasic Combined Oral Contraceptive (COC) Containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2), Compared to a Monophasic COC Containing 3 mg Drospirenone (DRSP) and 30 µg Ethinyl Estradiol (EE)
Brief Title: Efficacy and Safety Study of the Combined Oral Contraceptive NOMAC-E2 Compared to a COC Containing DRSP/EE (292002)(P05722)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05722; 292002
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOMAC-E2 (Experimental): Nomegestrol Acetate (NOMAC) and Estradiol (E2), 2.5 mg NOMAC and 1.5 mg E2 monophasic combined oral contraceptive
  Interventions: Drug: NOMAC-E2
- DRSP-EE (Active Comparator): Drospirenone (DRSP) and Ethinyl Estradiol (EE), 3 mg DRSP and 30 mcg EE monophasic combined oral contraceptive
  Interventions: Drug: DRSP-EE

INTERVENTIONS:
Drug: NOMAC-E2 — Nomegestrol Acetate and Estradiol Tablets, 2.5 mg NOMAC and 1.5 mg E2 taken once daily from Day 1 of menstrual period up to and including Day 28 for 13 consecutive 28-day menstrual cycles (1 year).
  Other Names: SCH900121; ORG10486-ORG2317
  Arms: NOMAC-E2
Drug: DRSP-EE — Drospirenone and Ethinyl Estradiol Tablets, 3 mg DRSP and 30 mcg EE taken once daily from Day 1 of menstrual period up to and including Day 28 for 13 consecutive 28-day menstrual cycles (1 year).
  Other Names: Yasmin
  Arms: DRSP-EE

SUMMARY:
The primary purpose of this study is to assess contraceptive efficacy, vaginal bleeding patterns (cycle control), general safety and acceptability of the nomegestrol acetate-estradiol (NOMAC-E2) combined oral contraceptive (COC) in a large group of women aged 18-50 years.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women, at risk for pregnancy and not planning to use condoms;
* Women in need for contraception and willing to use an oral contraceptive (OC) for 12 months (13 cycles);
* At least 18 but not older than 50 years of age at the time of screening;
* Body mass index >=17 and <=35;
* Good physical and mental health;
* Willing to give informed consent in writing.

Exclusion Criteria:

* Contraindications for contraceptive steroids
* In accordance with the Summary of Product Characteristics (SmPC)/Package Insert of DRSP-EE, additional contraindications related to the antimineralocorticoid activity of drospirenone (conditions that predispose to hyperkalemia):
* Renal insufficiency;
* Hepatic dysfunction;
* Adrenal insufficiency.
* An abnormal cervical smear (i.e.: dysplasia, cervical intraepithelial neoplasia [CIN], squamous intraepithelial lesion [SIL], carcinoma in situ, invasive carcinoma) at screening;
* Clinically relevant abnormal laboratory result at screening as judged by the investigator;
* Use of an injectable hormonal method of contraception; within 6 months of an injection with a 3-month duration, within 4 months of an injection with a 2-month duration, within 2 months of an injection with a 1-month duration;
* Before spontaneous menstruation has occurred following a delivery or abortion;
* Breastfeeding or within 2 months after stopping breastfeeding prior to the start of trial medication;
* Present use or use within 2 months prior to the start of the trial medication of the following drugs: phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, sex steroids (other than pre- and posttreatment contraceptive method) and herbal remedies containing Hypericum perforatum (St John's Wort);
* Administration of investigational drugs and/or participation in another clinical trial within 2 months prior to the start of the trial medication or during the trial period.
* Subjects with a diagnosis of the endometrial biopsy such as hyperplasia, atypical hyperplasia, carcinoma or any other abnormality judged clinically relevant by the investigator (This is applicable only for the subjects participating in the endometrial biopsy substudy).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2281 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

REFERENCES:
- [Derived] Witjes H, Creinin MD, Sundstrom-Poromaa I, Martin Nguyen A, Korver T. Comparative analysis of the effects of nomegestrol acetate/17 beta-estradiol and drospirenone/ethinylestradiol on premenstrual and menstrual symptoms and dysmenorrhea. Eur J Contracept Reprod Health Care. 2015;20(4):296-307. doi: 10.3109/13625187.2015.1016154. Epub 2015 Feb 25. PMID 25712537
- [Derived] Westhoff C, Kaunitz AM, Korver T, Sommer W, Bahamondes L, Darney P, Verhoeven C. Efficacy, safety, and tolerability of a monophasic oral contraceptive containing nomegestrol acetate and 17beta-estradiol: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):989-99. doi: 10.1097/AOG.0b013e318250c3a0. PMID 22525910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants from North America and South America
Pre-assignment Details: In total, 2281 participants were randomized (NOMAC-E2 n=1710; DRSP-EE n=571) but 2220 participants were treated (NOMAC-E2 n=1666; DRSP-EE n=554).
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
- DRSP-EE: Monophasic COC tablets containing 3 mg Drospirenone (DRSP) and 30 mcg Ethinyl Estradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
Period: Overall Study
Arm/Group | NOMAC-E2 | DRSP-EE
Started | 1666 | 554
Completed | 988 | 344
Not Completed | 678 | 210
Not completed — Adverse event/serious adverse event | 289 | 56
Not completed — Pre-treatment (serious) adverse event | 1 | 0
Not completed — Withdrawal of informed consent | 111 | 36
Not completed — Pregnancy | 15 | 5
Not completed — Pregnancy wish | 17 | 6
Not completed — Lost to Follow-up | 175 | 73
Not completed — Other reason | 70 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 | DRSP-EE | Total
Number analyzed (Participants) | 1666 | 554 | 2220
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (7.2) | 27.8 (7.0) | 27.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1666 | 554 | 2220
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of In-treatment Pregnancies (With +2 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: In-treatment pregnancies were pregnancies with an estimated date of conception from the day of first intake of trial medication up to and including the day of last (active or placebo) intake of trial medication extended with a maximum of two days. Each 13 cycles (28 days per cycle) of exposure constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 women years) that the women were under risk of becoming pregnant.
Time Frame: 1 year (13 cycles)
Population: The "restricted ITT" set included all participants treated except for 27 nonpregnant participants whose exposure was excluded due to limited credibility of diary data, & also excluded nonpregnant participants without >= 1 cycle expected to be at risk for pregnancy (with recorded use of condoms or w/o sexual intercourse, based on e-diary data).
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1370 | 444
Number analyzed (woman years (rounded to nearest integer)) | 684 | 233
Pregnancies per 100 woman years
  Overall group | 1.754 [0.9061 to 3.0632] | 3.005 [1.2082 to 6.1917]
  =<35 years old (n=1158; n=378) | 1.963 [0.9798 to 3.5119] | 3.092 [1.1347 to 6.7299]
  >35 years old (n=212; n=66) | 0.807 [0.0204 to 4.4977] | 2.572 [0.0651 to 14.33]

2. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding/Spotting
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding/spotting was defined as any episode that occurred during the "expected non-bleeding period" that was neither an early nor a continued withdrawal bleeding. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants with evaluable cycles.
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
participants
  Cycle 1 (n=1202 NOMAC-E2; n=398 DRSP-EE) | 370 | 84
  Cycle 2 (n=950 NOMAC-E2; n=308 DRSP-EE) | 243 | 55
  Cycle 3 (n=812 NOMAC-E2; n=256 DRSP-EE) | 196 | 40
  Cycle 4 (n=739 NOMAC-E2; n=236 DRSP-EE) | 152 | 34
  Cycle 5 (n=671 NOMAC-E2; n=229 DRSP-EE) | 139 | 29
  Cycle 6 (n=628 NOMAC-E2; n=207 DRSP-EE) | 125 | 18
  Cycle 7 (n=565 NOMAC-E2; n=196 DRSP-EE) | 104 | 25
  Cycle 8 (n=543 NOMAC-E2; n=189 DRSP-EE) | 97 | 23
  Cycle 9 (n=507 NOMAC-E2; n=173 DRSP-EE) | 85 | 30
  Cycle 10 (n=491 NOMAC-E2; n=170 DRSP-EE) | 93 | 29
  Cycle 11 (n=456 NOMAC-E2; n=160 DRSP-EE) | 83 | 27
  Cycle 12 (n=428 NOMAC-E2; n=152 DRSP-EE) | 70 | 15
  Cycle 13 (n=383 NOMAC-E2; n=133 DRSP-EE) | 62 | 20

3. Primary Outcome: Number of In-treatment Pregnancies (With +14 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: In-treatment pregnancies were pregnancies with an estimated date of conception from the day of first intake of trial medication up to and including the day of last (active or placebo) intake of trial medication extended with a period of 14 days. Each 13 cycles (28 days per cycle) of exposure constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 women years) that the women were under risk of becoming pregnant.
Time Frame: 1 year (13 cycles)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1370 | 444
Number analyzed (woman years (rounded to nearest integer)) | 684 | 233
Pregnancies per 100 woman years
  Overall group | 2.192 [1.2268 to 3.6154] | 4.293 [2.0587 to 7.8951]
  =<35 years old (n=1158; n=378) | 2.498 [1.3657 to 4.1913] | 4.638 [2.1208 to 8.8042]
  >35 years old (n=212; n=66) | 0.807 [0.0204 to 4.4977] | 2.572 [0.0651 to 14.33]

4. Secondary Outcome: Number of Participants With an Occurrence of Absence of Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Absence of withdrawal bleeding was defined as no bleeding/spotting episode that began during or continued into the "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
participants
  Cycle 1 (n=1202 NOMAC-E2; n=398 DRSP-EE) | 216 | 23
  Cycle 2 (n=950 NOMAC-E2; n=308 DRSP-EE) | 167 | 15
  Cycle 3 (n=812 NOMAC-E2; n=256 DRSP-EE) | 178 | 15
  Cycle 4 (n=739 NOMAC-E2; n=236 DRSP-EE) | 184 | 16
  Cycle 5 (n=671 NOMAC-E2; n=229 DRSP-EE) | 169 | 13
  Cycle 6 (n=628 NOMAC-E2; n=207 DRSP-EE) | 166 | 9
  Cycle 7 (n=565 NOMAC-E2; n=196 DRSP-EE) | 139 | 13
  Cycle 8 (n=543 NOMAC-E2; n=189 DRSP-EE) | 152 | 16
  Cycle 9 (n=507 NOMAC-E2; n=173 DRSP-EE) | 151 | 8
  Cycle 10 (n=491 NOMAC-E2; n=170 DRSP-EE) | 147 | 8
  Cycle 11 (n=456 NOMAC-E2; n=160 DRSP-EE) | 156 | 6
  Cycle 12 (n=428 NOMAC-E2; n=152 DRSP-EE) | 141 | 10
  Cycle 13 (n=383 NOMAC-E2; n=133 DRSP-EE) | 187 | 7

5. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding was defined as any bleeding episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding.
  Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
participants
  Cycle 1 (n=1202 NOMAC-E2; n=398 DRSP-EE) | 100 | 19
  Cycle 2 (n=950 NOMAC-E2; n=308 DRSP-EE) | 47 | 5
  Cycle 3 (n=812 NOMAC-E2; n=256 DRSP-EE) | 43 | 5
  Cycle 4 (n=739 NOMAC-E2; n=236 DRSP-EE) | 39 | 7
  Cycle 5 (n=671 NOMAC-E2; n=229 DRSP-EE) | 30 | 4
  Cycle 6 (n=628 NOMAC-E2; n=207 DRSP-EE) | 29 | 4
  Cycle 7 (n=565 NOMAC-E2; n=196 DRSP-EE) | 31 | 5
  Cycle 8 (n=543 NOMAC-E2; n=189 DRSP-EE) | 25 | 5
  Cycle 9 (n=507 NOMAC-E2; n=173 DRSP-EE) | 24 | 7
  Cycle 10 (n=491 NOMAC-E2; n=170 DRSP-EE) | 27 | 9
  Cycle 11 (n=456 NOMAC-E2; n=160 DRSP-EE) | 19 | 5
  Cycle 12 (n=428 NOMAC-E2; n=152 DRSP-EE) | 16 | 3
  Cycle 13 (n=383 NOMAC-E2; n=133 DRSP-EE) | 16 | 2

6. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Spotting (Spotting Only)
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough spotting was defined as any spotting episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding.
  Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
participants
  Cycle 1 (n=1202 NOMAC-E2; n=398 DRSP-EE) | 306 | 72
  Cycle 2 (n=950 NOMAC-E2; n=308 DRSP-EE) | 211 | 50
  Cycle 3 (n=812 NOMAC-E2; n=256 DRSP-EE) | 168 | 36
  Cycle 4 (n=739 NOMAC-E2; n=236 DRSP-EE) | 126 | 30
  Cycle 5 (n=671 NOMAC-E2; n=229 DRSP-EE) | 114 | 25
  Cycle 6 (n=628 NOMAC-E2; n=207 DRSP-EE) | 102 | 16
  Cycle 7 (n=565 NOMAC-E2; n=196 DRSP-EE) | 85 | 20
  Cycle 8 (n=543 NOMAC-E2; n=189 DRSP-EE) | 78 | 18
  Cycle 9 (n=507 NOMAC-E2; n=173 DRSP-EE) | 64 | 23
  Cycle 10 (n=491 NOMAC-E2; n=170 DRSP-EE) | 71 | 21
  Cycle 11 (n=456 NOMAC-E2; n=160 DRSP-EE) | 67 | 22
  Cycle 12 (n=428 NOMAC-E2; n=152 DRSP-EE) | 59 | 12
  Cycle 13 (n=383 NOMAC-E2; n=133 DRSP-EE) | 46 | 18

7. Secondary Outcome: Number of Participants With an Occurrence of Early Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Early withdrawal bleeding was defined as any withdrawal bleeding that started before the current "expected bleeding period".
  Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
participants
  Cycle 1 (n=1202 NOMAC-E2; n=398 DRSP-EE) | 175 | 46
  Cycle 2 (n=950 NOMAC-E2; n=308 DRSP-EE) | 68 | 14
  Cycle 3 (n=812 NOMAC-E2; n=256 DRSP-EE) | 66 | 24
  Cycle 4 (n=739 NOMAC-E2; n=236 DRSP-EE) | 48 | 9
  Cycle 5 (n=671 NOMAC-E2; n=229 DRSP-EE) | 36 | 11
  Cycle 6 (n=628 NOMAC-E2; n=207 DRSP-EE) | 28 | 11
  Cycle 7 (n=565 NOMAC-E2; n=196 DRSP-EE) | 22 | 11
  Cycle 8 (n=543 NOMAC-E2; n=189 DRSP-EE) | 29 | 13
  Cycle 9 (n=507 NOMAC-E2; n=173 DRSP-EE) | 17 | 9
  Cycle 10 (n=491 NOMAC-E2; n=170 DRSP-EE) | 27 | 13
  Cycle 11 (n=456 NOMAC-E2; n=160 DRSP-EE) | 17 | 7
  Cycle 12 (n=428 NOMAC-E2; n=152 DRSP-EE) | 10 | 6
  Cycle 13 (n=383 NOMAC-E2; n=133 DRSP-EE) | 9 | 6

8. Secondary Outcome: Number of Participants With an Occurrence of Continued Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Continued withdrawal bleeding was defined as any withdrawal bleeding that continued into the "expected non-bleeding period" of the next cycle.
  Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 12 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
Measure: Number; unit: participants
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
  n= number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
- DRSP-EE: Monophasic COC tablets containing 3 mg Drospirenone (DRSP) and 30 mcg Ethinyl Estradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
  n= number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
participants
  Cycle 1 (n=1179 NOMAC-E2; n=393 DRSP-EE) | 367 | 216
  Cycle 2 (n=939 NOMAC-E2; n=304 DRSP-EE) | 309 | 174
  Cycle 3 (n=794 NOMAC-E2; n=254 DRSP-EE) | 225 | 149
  Cycle 4 (n=730 NOMAC-E2; n=235 DRSP-EE) | 192 | 145
  Cycle 5 (n=659 NOMAC-E2; n=227 DRSP-EE) | 171 | 135
  Cycle 6 (n=617 NOMAC-E2; n=207 DRSP-EE) | 149 | 122
  Cycle 7 (n=555 NOMAC-E2; n=194 DRSP-EE) | 142 | 111
  Cycle 8 (n=540 NOMAC-E2; n=188 DRSP-EE) | 128 | 107
  Cycle 9 (n=503 NOMAC-E2; n=171 DRSP-EE) | 116 | 106
  Cycle 10 (n=486 NOMAC-E2; n=169 DRSP-EE) | 121 | 95
  Cycle 11 (n=455 NOMAC-E2; n=159 DRSP-EE) | 90 | 94
  Cycle 12 (n=421 NOMAC-E2; n=149 DRSP-EE) | 95 | 78

9. Secondary Outcome: Average Number of Breakthrough Bleeding/Spotting Days
Description: as for outcome 2
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had breakthrough bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
days
  Cycle 1 (n=370 NOMAC-E2; n=84 DRSP-EE) | 4.5 (3.6) | 4.0 (2.9)
  Cycle 2 (n=243 NOMAC-E2; n=55 DRSP-EE) | 3.5 (2.7) | 2.7 (2.3)
  Cycle 3 (n=196 NOMAC-E2; n=40 DRSP-EE) | 3.2 (2.5) | 2.6 (2.0)
  Cycle 4 (n=152 NOMAC-E2; n=34 DRSP-EE) | 3.5 (2.7) | 3.2 (2.5)
  Cycle 5 (n=139 NOMAC-E2; n=29 DRSP-EE) | 3.6 (3.0) | 2.6 (2.1)
  Cycle 6 (n=125 NOMAC-E2; n=18 DRSP-EE) | 3.2 (2.7) | 3.0 (1.7)
  Cycle 7 (n=104 NOMAC-E2; n=25 DRSP-EE) | 3.9 (2.9) | 2.9 (2.0)
  Cycle 8 (n=97 NOMAC-E2; n=23 DRSP-EE) | 3.4 (2.4) | 2.6 (2.4)
  Cycle 9 (n=85 NOMAC-E2; n=30 DRSP-EE) | 3.5 (3.2) | 3.2 (2.2)
  Cycle 10 (n=93 NOMAC-E2; n=29 DRSP-EE) | 2.6 (2.1) | 3.2 (2.1)
  Cycle 11 (n=83 NOMAC-E2; n=27 DRSP-EE) | 3.6 (2.5) | 2.9 (2.0)
  Cycle 12 (n=70 NOMAC-E2; n=15 DRSP-EE) | 2.9 (2.4) | 3.1 (2.9)
  Cycle 13 (n=62 NOMAC-E2; n=20 DRSP-EE) | 2.8 (2.2) | 3.0 (1.9)

10. Secondary Outcome: Average Number of Withdrawal Bleeding/Spotting Days
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Withdrawal bleeding was defined as bleeding/spotting episode that started during or continued into the "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had withdrawal bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1312 | 436
days
  Cycle 1 (n=986 NOMAC-E2; n=375 DRSP-EE) | 5.7 (5.0) | 6.0 (3.5)
  Cycle 2 (n=783 NOMAC-E2; n=293 DRSP-EE) | 5.0 (4.6) | 6.2 (17.1)
  Cycle 3 (n=634 NOMAC-E2; n=241 DRSP-EE) | 4.8 (4.4) | 6.6 (18.9)
  Cycle 4 (n=555 NOMAC-E2; n=220 DRSP-EE) | 4.5 (2.9) | 6.5 (19.8)
  Cycle 5 (n=502 NOMAC-E2; n=216 DRSP-EE) | 4.5 (3.5) | 6.6 (19.9)
  Cycle 6 (n=462 NOMAC-E2; n=198 DRSP-EE) | 4.1 (2.5) | 6.6 (20.8)
  Cycle 7 (n=426 NOMAC-E2; n=183 DRSP-EE) | 4.2 (3.4) | 6.5 (21.6)
  Cycle 8 (n=391 NOMAC-E2; n=173 DRSP-EE) | 4.1 (2.4) | 6.8 (22.3)
  Cycle 9 (n=356 NOMAC-E2; n=165 DRSP-EE) | 3.9 (2.2) | 6.9 (22.8)
  Cycle 10 (n=344 NOMAC-E2; n=162 DRSP-EE) | 4.2 (2.8) | 6.8 (23.0)
  Cycle 11 (n=300 NOMAC-E2; n=154 DRSP-EE) | 3.8 (1.9) | 6.8 (23.6)
  Cycle 12 (n=287 NOMAC-E2; n=142 DRSP-EE) | 3.8 (2.5) | 6.9 (24.6)
  Cycle 13 (n=196 NOMAC-E2; n=126 DRSP-EE) | 2.8 (2.3) | 4.3 (1.6)

ADVERSE EVENTS:
Arm/Group | NOMAC-E2 | DRSP-EE
Serious Adverse Events (participants affected / at risk) | 32/1666 | 6/554
Other Adverse Events (participants affected / at risk) | 720/1666 | 162/554
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=1666) | DRSP-EE (N=554)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Venous angioma of brain (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumor of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Degeneration of uterine fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (2) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Breast cosmetic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=1666) | DRSP-EE (N=554)
Weight increased (Investigations) | 210 (215) | 38 (38)
Headache (Nervous system disorders) | 121 (162) | 46 (69)
Cervical dysplasia (Reproductive system and breast disorders) | 77 (78) | 34 (35)
Metrorrhagia (Reproductive system and breast disorders) | 102 (120) | 17 (18)
Withdrawal bleeding irregular (Reproductive system and breast disorders) | 154 (293) | 3 (6)
Acne (Skin and subcutaneous tissue disorders) | 327 (390) | 60 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the SPONSOR. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the SPONSOR, at least six weeks ahead of estimated publication or presentation, for consent, which shall not be withheld unreasonably.